CLINICAL TRIAL: NCT03402724
Title: Long Term Clinical and Echographic Follow Up After TAVI: A Pro-spective Cohort Study.
Brief Title: Long-term Clinical and Echographic Follow-up (More Than 4 Years) After TAVI.
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF7570
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Severe and Symptomatic Aortic Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: echographic — Patients are called for an echographic evaluation in the implanting center in case of the usual care

SUMMARY:
Transcatheter Aortic Valve Implantation (TAVI) is became the gold-standard therapy for patients with severe and symptomatic aortic stenosis with high operative risk or not suitable for surgery.

All studies assessed TAVI showed excellent results at short and mid-term follow-up. The current and future development of the devices predict an extension of indications to "intermediate-risk" and younger patients.

Therefore, long-term evaluation of these valves is a priority to determine their durability.

However, standardized echographic follow-up of patients implanted with TAVI is lacking.

Indeed, there was not consensual definition of TAVI degeneration until now. Recently, European Society of Cardiology published echographic criteria to precise and standardized TAVI deterioration based on simple hemodynamic and morphological criteria.

In addition, very few studies have been interested in monitoring more than 5 years of these devices.

Finally, nowadays we did not know if TAVI evolution is the same as surgical bioprosthesis.

DETAILED DESCRIPTION:
Transcatheter Aortic Valve Implantation (TAVI) is became the gold-standard therapy for patients with severe and symptomatic aortic stenosis with high operative risk or not suitable for surgery.

All studies assessed TAVI showed excellent results at short and mid-term follow-up. The current and future development of the devices predict an extension of indications to "intermediate-risk" and younger patients.

Therefore, long-term evaluation of these valves is a priority to determine their durability.

Clinical outcomes of these patients are well documented by large registers. Thus, FRANCE 2 registry studying more than 3000 patients realized in 34 French centers showed at 30 days a rate of death of 9.7%, and incidence of stroke of 3.4%. SOURCE registries studied more than 5000 patients in Europe and United-States with three generations of TAVI. All-cause mortality at 1 year was respectively 23.9%, 19.4% and 11.7% in SOURCE, SOURCE XT (Sapien XT) and SOURCE 3 (Sapien 3).

However, standardized echographic follow-up of patients implanted with TAVI is lacking.

Indeed, there was not consensual definition of TAVI degeneration until now. Recently, European Society of Cardiology published echographic criteria to precise and standardized TAVI deterioration based on simple hemodynamic and morphological criteria.

In addition, very few studies have been interested in monitoring more than 5 years of these devices.

Finally, nowadays the investigator did not know if TAVI evolution is the same as surgical bioprosthesis.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients admitted from February 2010 to December 2014 at the University Hospital of Montpellier for the implantation of TAVI will be included for TAVI Edwards.
* Male or non-pregnant female ≥ 18 years without superior limit of age for TAVI, indicated for severe and sympto-matic aortic valve stenosis, defined according to the guidelines (1), with high-surgical risk or not suitable for surgery, and after Heart Team decision.
* Informed consent obtained at enrolment into the study

Exclusion criteria:

* Inability to give informed consent or high likelihood of being unavailable for follow-up
* Patients died during the implantation and within one year after implantation will be excluded because of impossibil-ity of follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted from February 2010 to December 2014 at the University Hospital of Montpellier for the implantation of TAVI will be included for TAVI Edwards.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
echographic follow-up | 1 day
  - echographic follow-up more than 4 years of TAVI implanted in CHU of Montpellier, using new echographic criteria defined by European Socizty of Cardiology

CONTACTS AND LOCATIONS:
Overall Officials: Florence LECLERCQ, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC